CLINICAL TRIAL: NCT05709665
Title: Incidence and Special Informations From Patients of the Out- and in Hospital Cardiac Arrest at a Tertiary Hospital in Germany
Brief Title: Incidence of the Out- and in Hospital Cardiac Arrest at a Tertiary Hospital in Germany
Acronym: ProseCPR
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Johannes Gutenberg University Mainz (Other)
Responsible Party: Principal Investigator, Marc Kriege, MD, Principal Investigator, Johannes Gutenberg University Mainz
Other Study IDs: JohannesGUC
Record Dates: First submitted 2023-01-24; First posted 2023-02-02 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Resuscitation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Out-of-hospital cardiac arrest: Patient characteristics; Rescue time intervals; Time to eCPR Decision during high quality CPR;
  Interventions: Other: Time to Decision for eCPR
- In-hospital cardiac arrest: Patient characteristics; Emergency team time intervals; Time to eCPR Decision during high quality CPR;
  Interventions: Other: Time to Decision for eCPR

INTERVENTIONS:
Other: Time to Decision for eCPR — We evaluate during high quality CPR the time for decision for eCPR
  Other Names: Pros eCPR

SUMMARY:
Incidence of the background information, incidence and special characteristics of out- and in-hospital cardiac arrest at a tertiary hospital in Germany.

DETAILED DESCRIPTION:
To evaluate background information for planning a eCPR Program at a tertiary hospital, the investigators planned a prospective study of every out- and in-hospital cardiac arrest.

ELIGIBILITY:
Inclusion Criteria:

* All patients with a cardiac arrest

Exclusion Criteria:

* not complete fill out evaluation forms

Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: All cardiac arrest patients at a tertiary hospital
Sampling Method: Non-Probability Sample
Enrollment: 80 (Estimated)
Dates: Start 2023-01-11 (Actual); Primary Completion 2023-07-11 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
Time to eCPR Decision during high quality CPR | < 10 Minutes
  After established high quality CPR, we evaluate the time of decision for eCPR

SECONDARY OUTCOMES:
Patient characteristics | < 10 Minutes
  Age, BMI, comorbidity, contraindications for ECMO
Rescue/Emergency team time intervals | < 60 Minutes
  Time to Achievement at the patient; Time for transport

CONTACTS AND LOCATIONS:
Overall Officials: Marc Kriege, MD, Principal Investigator — University Medical Center Mainz
Locations (1):
- Department of Anesthesiology,Prof. C. Werner, Universitätsmedizin of the JG University, Mainz, Rhineland-Palatinate, Germany

IPD SHARING:
Plan to Share IPD: No